CLINICAL TRIAL: NCT00063869
Title: A Double-blind, Parallel, Placebo-controlled, Randomized Study of the Efficacy and Safety of Etanercept in Patients With Idiopathic Pulmonary Fibrosis.
Brief Title: Study Evaluating the Safety and Efficacy of Etanercept in Patients With Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0881A4-203
Record Dates: First submitted 2003-07-07; First posted 2003-07-09 (Estimated); Last update posted 2009-09-04 (Estimated); Status verified 2009-09

CONDITIONS: Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis; Fibrosis, Pulmonary; Pulmonary Fibroses; Fibroses, Pulmonary
MeSH Terms: conditions — Pulmonary Fibrosis; Idiopathic Pulmonary Fibrosis | interventions — Etanercept

INTERVENTIONS:
Drug: Etanercept

SUMMARY:
The objective of the study is to evaluate the safety and efficacy of etanercept in comparison with placebo in a double-blind, parallel, randomized fashion in subjects with idiopathic pulmonary fibrosis (IPF) who failed previous therapy. The treatment period will be up to 1 year. The primary objective is evaluation of safety and efficacy. Secondary: The secondary objective is to evaluate quality of life (QoL) and pharmacokinetics (PK).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IPF based on American Thoracic Society (ATS) guidelines

Exclusion Criteria:

* Subjects with end-stage
* Previous treatment with etanercept or other TNF antagonists (eg, a TNF monoclonal antibody or a soluble TNF-receptor)
* Receipt of any investigational drug or biological agent within 4 weeks of screening visit

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Raghu G, Brown KK, Costabel U, Cottin V, du Bois RM, Lasky JA, Thomeer M, Utz JP, Khandker RK, McDermott L, Fatenejad S. Treatment of idiopathic pulmonary fibrosis with etanercept: an exploratory, placebo-controlled trial. Am J Respir Crit Care Med. 2008 Nov 1;178(9):948-55. doi: 10.1164/rccm.200709-1446OC. Epub 2008 Jul 31. PMID 18669816